CLINICAL TRIAL: NCT06819943
Title: Effectiveness of Platform-Based Lateralization Therapy in Reducing Interface Pressure Between The Patient And The Support Surface
Acronym: PREVENT-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcelo Britto Passos Amato, MD PHD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 73162823.2.0000.0068
Record Dates: First submitted 2025-01-22; First posted 2025-02-11 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Insufficiency; Pressure Injury; Intensive Care Medicine; ARDS
Keywords: Continuous Lateral Rotation Therapy; Rotation Therapy
MeSH Terms: conditions — Respiratory Insufficiency; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Crossover study with Latin Square allocation. All participants are exposed to both automated lateral tilt and the supine reference position, in a balanced order, with washout periods between conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Automated Lateral Rotation Therapy (Experimental): Experimental positioning protocol with automated lateral rotation. After allocation, each participant is assigned to an initial lateralization side (right or left) and an initial head-of-bed elevation (10 or 30 degrees). The protocol begins with arterial blood gas sampling in the supine position. Lateralization follows a fixed sequence of 15 and 30 degrees, held for 10 minutes each, first on the assigned side and then on the opposite side. Each position is separated by a 10-minute washout period in the supine position with the same head-of-bed elevation. After completing this sequence, the participant returns to the supine position, and the second head-of-bed elevation (the one not initially assigned) is applied, repeating the same sequence starting again from the same lateralization side assigned initially. At the end of the protocol, a post-protocol arterial blood gas is collected. All positions are maintained for 10 minutes each.
  Interventions: Procedure: Automated Lateral Rotation Therapy

INTERVENTIONS:
Procedure: Automated Lateral Rotation Therapy — Platform-based automated lateral tilt system integrated into the Linet Multicare bed, which allows the entire bed platform to be tilted laterally up to 30 degrees along the axial axis, either manually or automatically. The system includes Continuous Low Pressure (CLP) mode, which automatically redistributes pressure to maintain low interface pressure, and Microclimate Management (MCM) to control moisture and heat at the skin interface. The intervention is designed to redistribute interface pressure as a preventive strategy against pressure injuries in critically ill patients.

SUMMARY:
Pressure injury (PI) is characterized as damage to the skin and/or underlying tissues resulting from sustained pressure or a combination of pressure and shear forces between the patient and the support surface. Prolonged pressure is a well-established risk factor in the development of PIs. Frequent repositioning and routine patient care have been recognized for decades as integral components of PI prevention and treatment protocols.

The duration of interface pressure is as critical as its magnitude. When interface pressure exceeds the mean capillary blood pressure, blood flow can be compromised, leading to ischemia in affected areas, which may progress to necrosis if sustained over time. Furthermore, it is widely accepted in the literature that tissue becomes at risk when interface pressure exceeds 30 to 32 mmHg.

In this context, continuous lateral rotation therapy (CLRT) offers a potential alternative for managing critically ill patients. CLRT involves continuous mechanical rotation of the patient in the lateral plane. However, its effects on skin integrity remain poorly understood. Despite the rationale behind and widespread recommendation of repositioning, the lack of robust evaluations on how repositioning impacts interface pressure creates uncertainty, underscoring the need for high-quality trials to assess different strategies for implementation.

Although lateralization is a pragmatic strategy for preventing pressure injuries, its use in critically ill patients requires an integrated assessment of respiratory, hemodynamic, and gastroesophageal effects. Therefore, this study proposes an innovative approach by evaluating, for the first time, the effectiveness of automated postural change with simultaneous monitoring of tissue integrity, pulmonary function, cardiovascular stability, and gastroesophageal protection. The aim is to optimize pressure injury prevention, improve pulmonary mechanics, ensure hemodynamic stability, and preserve gastroesophageal safety in critically ill patients.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effectiveness of Automated Lateral Rotation Therapy in reducing interface pressure between the patient and the support surface, considering different head-of-bed elevations, in mechanically ventilated patients. This is a multidimensional approach, assessing the effects on respiratory, hemodynamic, and gastroesophageal parameters.

This is a single-center, intra-individual crossover randomized clinical trial, using a Latin square allocation model, conducted in an intensive care unit.

The study will compare the effects of automated platform lateralization at 15 degrees and 30 degrees, combined with a 10-degree head-of-bed elevation, to the supine position with a 30-degree head-of-bed elevation, focusing on the reduction of interface pressure. Lateral tilting will be performed to both sides (right and left) according to prior randomization. Each position will be maintained for 10 minutes, followed by a 10-minute washout period in the supine position before transitioning to the next condition.

Additionally, after completing the crossover assessments, a subgroup of six patients will undergo an extended monitoring phase. In this step, the lateralized position at 30 degrees with a 30-degree head-of-bed elevation will be maintained for two continuous hours on each side (right and left) to assess the temporal evolution of interface pressure, determining whether pressure values remain stable or tend to increase over time.

The intervention will be conducted using the Linet Multicare bed, equipped with the Symbioso mattress, which features Continuous Low Pressure (CLP) and Microclimate Management (MCM) modes. This system enables manual or automated lateral tilting of the entire bed platform up to 30 degrees on the axial axis. The CLP mode provides automatic, continuous low-pressure redistribution, minimizing interface pressures regardless of weight distribution or patient movement. The MCM mode includes a vapor-impermeable cover that reduces skin moisture and heat, supporting skin integrity and preventing maceration.

Monitoring Procedures Interface pressure monitoring will be performed using the ForeSite Intelligent Surface (Xsensor, Canada), a sensor network embedded in a mattress cover composed of 6136 sensing cells distributed over an area of 762 by 1880 millimeters, with a spatial resolution of 31.75 millimeters. The system provides continuous pressure acquisition at 3 Hz, operating in the range of 5 to 200 mmHg (0.7 to 36.6 kPa), with an accuracy of plus or minus 2 mmHg. During the protocol, interface pressure will be monitored continuously with real-time visual feedback displayed on a bedside LCD monitor, allowing visualization of pressure redistribution throughout the interventions.

Pulmonary monitoring will be conducted using the ENLIGHT (Timpel, model 2100, Brazil), which utilizes a 32-electrode belt placed around the thorax at the mid-axillary line to provide real-time monitoring of ventilation distribution through electrical impedance tomography (EIT).

Hemodynamic monitoring will be performed using the FloTrac system coupled with the EV1000 platform (Edwards Lifesciences, Irvine, California, USA), connected to a peripheral arterial catheter, enabling continuous measurement of cardiac output, cardiac index, stroke volume, stroke volume variation, and blood pressure parameters.

Gastroesophageal pH monitoring will be carried out using the AL-4 pH monitoring system (ALACER, Brazil), which includes an antimony pH probe with an external reference electrode placed on the patient's thoracic skin to continuously measure esophageal pH levels.

Primary Hypothesis Automated Lateral Rotation Therapy promotes a reduction in interface pressure, assessed by peak pressure, mean pressure, and the absolute count of sensors recording pressure above 40 mmHg. Additionally, it is hypothesized that the extent of this reduction varies depending on the degree of lateral tilt and head-of-bed elevation, with lower degrees potentially being more effective for pressure redistribution.

Secondary Hypotheses Automated lateral positioning improves respiratory mechanics, contributing to better ventilation and oxygenation.

Adverse hemodynamic effects are minimized when using controlled tilt angles. Automated lateral rotation does not increase the incidence of gastroesophageal reflux.

Primary Outcome Reduction in peak pressure in the sacral region.

Secondary Outcomes Peak pressure mean pressure in the occipital, scapular, and calcaneal regions. Mean pressure in the sacral, occipital, scapular, and calcaneal regions. Number of sensors with pressure above 32, 40, and 60 mmHg in the sacral, occipital, scapular, and calcaneal regions.

Respiratory parameters including static compliance, driving pressure, oxygenation, and volumetric capnography.

Hemodynamic parameters including heart rate, blood pressure, cardiac output, cardiac index, stroke volume, and stroke volume variation.

Gastric pH variation during different positioning conditions. Adverse events including hypotension, accidental ventilator disconnection, respiratory discomfort, or significant gastroesophageal reflux.

Pre-intervention Procedures

Before starting the protocol, a standardized preparation process will be performed to ensure clinical stability, measurement accuracy, and consistency across all participants. The following procedures will be applied:

Closed-system suctioning to minimize secretion accumulation and avoid measurement artifacts.

Adjustment of ventilator settings in Volume-Controlled Ventilation (VCV) mode, using a square wave flow pattern. Respiratory rate (RR), inspiratory-to-expiratory ratio (I:E), fraction of inspired oxygen (FiO₂), and tidal volume (Vt) will be maintained according to baseline parameters.

Positive End-Expiratory Pressure (PEEP) will be maintained at the baseline value plus 2 cmH₂O during lateralization phases, to compensate for potential changes in thoracic mechanics and prevent derecruitment.

Placement of the interface pressure sensor (ForeSite PT, XSENSOR) will be performed by two trained professionals to ensure correct positioning, alignment, and reduction of artifacts.

Bed surface and sensor positioning will be inspected to eliminate any folds, misalignments, or sensor displacements that could interfere with pressure measurements.

The esophageal pH monitoring system will be zeroed and calibrated before each change in the head-of-bed elevation, ensuring accurate pH recording.

Proton pump inhibitor (PPI) administration will be rescheduled prior to the protocol, and the enteral feeding tube must be confirmed in a post-pyloric position, reducing the risk of reflux and interference with pH measurements.

ELIGIBILITY:
Inclusion Criteria

* Adult and elderly patients, aged 18 years or older;
* Patients under controlled or assisted mechanical ventilation, not yet eligible for weaning.

Exclusion Criteria

* Requirement of norepinephrine > 0.3 mcg/kg/min or mean arterial pressure < 60 mmHg, despite the use of vasopressor agents;
* Cardiac arrhythmias or bleeding leading to hemodynamic instability;
* Neurological diseases or symptoms;
* Spinal cord injury, such as paraplegia;
* Cardiac pacemaker dependence;
* Contraindications to hypercapnia, such as intracranial hypertension or acute coronary syndrome;
* Air leakage from chest drains, presence of pneumothorax or undrained subcutaneous emphysema;
* Presence of pre-existing pressure injuries in bony prominences (sacral, occipital, scapular, or calcaneal) at admission;
* Medical refusal to include the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Interface Pressure | Pressure measurements correspond to the mean value during the 10 minutes of each position, for both head-of-bed inclinations. In the extended monitoring phase, data are collected continuously for 2 hours on each side.
  The interface pressure will be measured from the pressure reading made by the XSensor. The average pressure, peak pressure, and median pressure will be used for each region of the body. In addition to the absolute count of pressure sensors that made a reading above 32, 40 and 60mmHg.

SECONDARY OUTCOMES:
Driving Pressure | Readings will be taken immediately before changing to the next position, after stabilization in each position, during the protocol.
  Driving Pressure (cmH2O) will be measured using the information provided by the EIT that uses the movement equation
End Expiratory Lung Volume | Readings will be taken immediately before changing to the next position, after stabilization in each position, during the protocol.
  Will be measured using the information provided by the Electrical Tomography Impedance
Ventilatory Distribution | Readings will be taken immediately before changing to the next position, after stabilization in each position, during the protocol.
  Will be measured using the information provided by the Electrical Tomography Impedance
Plateau Pressure | Readings will be taken immediately before changing to the next position, after stabilization in each position, during the protocol.
  Plateau Pressure( cmH2O) will be measured using the information provided by the EIT that uses the movement equation.
Esophageal reflux | It uses a pH probe that will be kept continuously during the protocol. The pH curve over time is analyzed offline using the software provided by ALACER.
  Measurement with pH meter probe from Alacer Biomédica.
Diastolic Blood Pressure | Readings will be taken immediately before changing to the next position, after stabilization in each position, during the protocol.
  The hemodynamics were assessed through Diastolic Blood Pressure using the multiparameter monitor DX-2020 (Dixtal, São Paulo, Brazil).
Mean Arterial Pressure | Readings will be taken immediately before changing to the next position, after stabilization in each position, during the protocol.
  The hemodynamics were assessed through Mean Artial Pressure using the multiparameter monitor DX-2020 (Dixtal, São Paulo, Brazil).
Systolic Blood Pressure | Readings will be taken immediately before changing to the next position, after stabilization in each position, during the protocol.
  The hemodynamics were assessed through Systolic Blood Pressure using the multiparameter monitor DX-2020 (Dixtal, São Paulo, Brazil).
Heart Rate | Readings will be taken immediately before changing to the next position, after stabilization in each position, during the protocol.
  The hemodynamics were assessed through Heart Rate using the multiparameter monitor DX-2020 (Dixtal, São Paulo, Brazil).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da Universidade São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miranda DR, Nap R, de Rijk A, Schaufeli W, Iapichino G; TISS Working Group. Therapeutic Intervention Scoring System. Nursing activities score. Crit Care Med. 2003 Feb;31(2):374-82. doi: 10.1097/01.CCM.0000045567.78801.CC. PMID 12576939
- [Background] Peterson MJ, Schwab W, van Oostrom JH, Gravenstein N, Caruso LJ. Effects of turning on skin-bed interface pressures in healthy adults. J Adv Nurs. 2010 Jul;66(7):1556-64. doi: 10.1111/j.1365-2648.2010.05292.x. Epub 2010 May 21. PMID 20497272
- [Background] Ayello EA, Braden B. How and why to do pressure ulcer risk assessment. Adv Skin Wound Care. 2002 May-Jun;15(3):125-31; quiz 132-33. doi: 10.1097/00129334-200205000-00008. PMID 12055446
- [Background] Bergstrom N, Braden BJ, Laguzza A, Holman V. The Braden Scale for Predicting Pressure Sore Risk. Nurs Res. 1987 Jul-Aug;36(4):205-10. PMID 3299278
- [Background] Anderson R, Kleiber C, Greiner J, Comried L, Zimmerman M. Interface pressure redistribution on skin during continuous lateral rotation therapy: A feasibility study. Heart Lung. 2016 May-Jun;45(3):237-43. doi: 10.1016/j.hrtlng.2016.02.003. Epub 2016 Mar 15. PMID 26992481